CLINICAL TRIAL: NCT07204327
Title: Effectiveness and Safety of Atezolizumab + Bevacizumab Plus Locoregional Therapies in Patients With Unresectable Hepatocellular Carcinoma in Real-world Clinical Practice
Brief Title: Atezolizumab Plus Bevacizumab Combined With Locoregional Therapies in Unresectable Hepatocellular Carcinoma (ISMIO-001)
Acronym: ISMIO001
Status: Active, not recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Center of Interventional Radiology and Vascular Surgery, Zhongda Hospital
Other Study IDs: CHANCE2510-ISMIO001
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Atezolizumab; Bevacizumab; Unresectable HCC; Locoregional Therapy; TACE; HAIC; TARE; Ablation; Real-world; HBV; Asia-Pacific

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- uHCC patients treated with Atezo+Bev plus LRT: Patients with unresectable hepatocellular carcinoma (uHCC) who received first-line atezolizumab plus bevacizumab (Atezo+Bev) in combination with at least one locoregional therapy (TACE, HAIC, TARE, ablation, or radiotherapy) within ±2 months of systemic therapy initiation, between October 28, 2020 and July 31, 2025.
  Interventions: Other: Atezo+Bev plus Locoregional Therapy

INTERVENTIONS:
Other: Atezo+Bev plus Locoregional Therapy — Patients received atezolizumab plus bevacizumab (Atezo+Bev) in combination with at least one locoregional therapy (transarterial chemoembolization [TACE], hepatic arterial infusion chemotherapy [HAIC], transarterial radioembolization [TARE], ablation, or radiotherapy) within ±2 months of systemic therapy initiation, in routine clinical practice.

SUMMARY:
This is a retrospective, multicenter, real-world cohort study designed to evaluate the effectiveness and safety of atezolizumab plus bevacizumab (Atezo+Bev) combined with various locoregional therapies (LRTs), including transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), transarterial radioembolization (TARE), ablation, and radiotherapy, in patients with unresectable hepatocellular carcinoma (uHCC). Approximately 1,136 patients treated between October 28, 2020 and October 31, 2025 will be included from about 35 sites across China and the Asia-Pacific region. The primary endpoint is overall survival (OS). Secondary endpoints include real-world progression-free survival (rwPFS), overall response rate (ORR), disease control rate (DCR), time to discontinuation (TTD), time to next treatment (TTNT), time to progression (TTP), and safety outcomes. Exploratory analyses will assess associations between baseline patient characteristics, treatment patterns, and clinical outcomes.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a major cause of cancer-related death worldwide, with a particularly high burden in China and the Asia-Pacific region, where chronic hepatitis B virus (HBV) infection is the predominant etiology. While atezolizumab plus bevacizumab (Atezo+Bev) has been established as the global first-line standard of care for unresectable HCC (uHCC), clinical trial populations were highly selective, excluding patients with impaired liver function or poor performance status, and the overall response rate remains limited at approximately 30%.

Locoregional therapies (LRTs) such as TACE, HAIC, TARE, ablation, and radiotherapy remain an integral part of uHCC management in the Asia-Pacific region, offering potential synergistic effects when combined with Atezo+Bev. However, there is a lack of robust real-world evidence describing the timing, sequencing, and outcomes of these combined strategies.

The ISMIO-001 study is designed as a retrospective, multicenter, real-world cohort study. Eligible patients must be ≥18 years old, diagnosed with uHCC, and treated with Atezo+Bev plus at least one LRT within ±2 months of Atezo+Bev initiation, between October 28, 2020 and July 31, 2025. The observation period will continue until October 31, 2025, with study completion anticipated by December 31, 2026.

The study will provide large-scale evidence on treatment patterns, overall survival, safety, and subgroup outcomes (e.g., by BCLC/CNLC stage, Child-Pugh class, ALBI grade, HBV vs. other etiologies). Findings will inform future clinical guidelines and support the optimization of treatment sequencing for uHCC in HBV-predominant populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at initiation of atezolizumab plus bevacizumab (Atezo+Bev)
* Histologically or radiologically confirmed unresectable hepatocellular carcinoma (uHCC) according to national guidelines
* Initiated first-line Atezo+Bev treatment between October 28, 2020 and July 31, 2025
* Received ≥1 locoregional therapy (TACE, HAIC, TARE, ablation, or radiotherapy) within ±2 months of Atezo+Bev initiation
* At least one follow-up record available after treatment initiation

Exclusion Criteria:

* Prior systemic therapy for HCC before Atezo+Bev initiation
* Concurrent participation in interventional clinical trials at baseline
* Diagnosis of other malignancies at baseline (except basal cell carcinoma of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable hepatocellular carcinoma (uHCC) treated in routine clinical practice across multiple centers in China and the Asia-Pacific region, receiving atezolizumab plus bevacizumab in combination with locoregional therapies.
Sampling Method: Non-Probability Sample
Enrollment: 1136 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 36 months (median follow-up period anticipated)
  Overall survival, defined as the time from initiation of atezolizumab plus bevacizumab treatment to death from any cause.

SECONDARY OUTCOMES:
Real-world Progression-Free Survival (rwPFS) | Up to 36 months
  Time from initiation of Atezo+Bev treatment to investigator-assessed disease progression (local progression, recurrence, new metastasis, or clinical progression) or death from any cause.
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with complete response (CR) or partial response (PR), as assessed by RECIST 1.1 and mRECIST criteria.
Disease Control Rate (DCR) | Up to 36 months
  Proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD ≥6 weeks), based on RECIST 1.1 or mRECIST.
Time to Treatment Discontinuation (TTD) | Up to 36 months
  Time from treatment initiation to discontinuation of Atezo+Bev for any reason.
Time to Next Treatment (TTNT) | Up to 36 months
  Time from initiation of Atezo+Bev to start of subsequent systemic therapy.
Time to Progression (TTP) | Up to 36 months
  Time from initiation of Atezo+Bev to first documentation of disease progression.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to 36 months
  Incidence and severity of all adverse events (AEs), treatment-related AEs (TRAEs), and adverse events of special interest (bleeding, hypertension, hepatic impairment, immune-related AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Yes, de-identified IPD may be shared upon reasonable request

DOCUMENTS (1):
  • Study Protocol (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT07204327/Prot_000.pdf